CLINICAL TRIAL: NCT03738306
Title: Mézières Method for "The Use of Self" in People With Low Back Pain. Mixed Study.
Brief Title: Mézières Method in People With Low Back Pain.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de la Sabana (Other)
Collaborators: Universidad Ramón Llull (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENF-26-2018
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mezieres Method (Experimental): The Mézières treatment has 3 postures that could be adapted to each patient, depending on his/her needs to correct variations in the dorsal curve and promote diaphragmatic breathing. The first objective was to recover extensibility of the hypertonic muscle groups and, in particular, those in the low back muscular chain. The time of tratment will be of 1 hour, two times a week, during 5 weeks.
  Interventions: Other: Mezieres Method
- Conventional Physiotherapy (Active Comparator): The treatment with conventional physiotherapy will include stretching of hamstrings, gluteus, (and others) hot pack, transcutaneous electrical nerve stimulation, ultrasound and some exercises of core performance.The time of treatment will be of 1 hour, two times a week, during 5 weeks.
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Mezieres Method — "The Mézières treatment have 3 postures that could be adapted to each patient, depending on his/her needs to correct variations in the dorsal curve and promote diaphragmatic breathing. The first objective was to recover extensibility of the hypertonic muscle groups and, in particular, those in the low back muscular chain: the paravertebral muscles and latissimus dorsi".
  Arms: Mezieres Method
Other: Conventional Physiotherapy — therapeutic exercise; physical agents
  Arms: Conventional Physiotherapy

SUMMARY:
The Mezieres method was born in France with the physiotherapist Francoiçe Mezieres, who in the middle of the previous century began a series of observations that led her to rediscover body characteristics to understand it in a revolutionary way. Among the most important contributions is the first description of muscle chains, from which different global physiotherapy techniques have emerged. The method also proposes a form of intercorporal relationship different from that used in classical physiotherapy and gives way for people who receive this treatment to improve their body disposition and make use of their body in a conscientious manner. From this, in the present study we try to understand this method as one of the ones that promotes the "Use of self". In addition to identifying other aspects related to the meaning of the corporal intersubjectivity for the physiotherapist and for the person being treated, looking for the subjective construction of effectiveness and determining the objective effectiveness by means of objective measurements of the body.

The present research project use a mix method, it aims quantify the bodily benefits when applying the method and understand from the subjectivity the implications for the self during the body activity of the Mezieres Method. The study will be mixed and in parallel with 82 people diagnosed with mechanical back pain. Three assessments will be made: one initial, one at the end of the intervention and one last follow-up six weeks after the end of the treatment. The tests to be used will assess pain, functional limitation related to low back pain, quality of life related to health, flexibility, range of motion and posture. For the intervention, participants will be divided into 2 groups, group one will receive Method Mézières and group two will receive conventional physiotherapy according to the protocols of a clinical institution in Bogotá. Parallel to the intervention, the participating individuals and physiotherapists will keep a field diary that will facilitate the understanding of the body experience by performing the method studied.

At the end of the study, it is intended to know the objective effectiveness by means of the comparison made in the two groups in the variables studied. In addition, an interpretation of the body experience is expected when performing the Mezieres Method in comparison with conventional physiotherapy. This interpretation of hermeneutic character will revolve around the theoretical construction of the "Use of self"; This concept is recognized as a technology of the self that will be pursued through the Mézières Method. By promoting the "Use of self" the person can recognize their body and appropriate what happens with their locomotor system, decreasing the symptoms of pain and improving the prognosis of care for people who have these symptoms.

ELIGIBILITY:
Inclusion Criteria:

* People with low back pain (LBP) (mechanical)
* people with LBP of at least three months
* people with LBP with a requirement from medicine to be treated by physiotherapy
* people with Roland Morris Questionnaire major to 4.

Exclusion Criteria:

* Anamnesis with red flags related with low back pain
* signs of lumbar pain associated with compression or radicular injury
* shortening of the lower limb or any mechanical modification that affects the lumbopelvic complex.
* post-surgery of the spine
* symptoms of depression or emotional risk factors that worsen the clinical

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Roland Morris Questionnaire | 5 weeks
  Self reported Disability related with low back pain, the score is 0- 24. It will be applied in the initial evaluation, after of five weeks of intervention and 6 weeks after of second evaluation.
Health Related Quality of Life | 5 weeks
  Questionnaire consist in twelve questions that e assessment difference health domains related with quality of life

SECONDARY OUTCOMES:
Posture | 5 weeks
  Alignment with gravity line. We Will take a photography, it will be analyzed in a ADIBAS software to identificate the alignment of the participant according to the line gravity.
Trunk Range of movement | 5 weeks
  The mobee digital goniometer is used to calculate the flexion and trunk extension angle

CONTACTS AND LOCATIONS:
Overall Officials: Margareth L Alfonso-Mora, Mg, Principal Investigator — Universiad de La Sabana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pellecchia MT, Grasso A, Biancardi LG, Squillante M, Bonavita V, Barone P. Physical therapy in Parkinson's disease: an open long-term rehabilitation trial. J Neurol. 2004 May;251(5):595-8. doi: 10.1007/s00415-004-0379-2. PMID 15164194
- [Background] Pepe L, Milani R, Di Trani M, Di Folco G, Lanna V, Solano L. A more global approach to musculoskeletal pain: expressive writing as an effective adjunct to physiotherapy. Psychol Health Med. 2014;19(6):687-97. doi: 10.1080/13548506.2013.859712. Epub 2013 Nov 20. PMID 24251961
- [Background] Valencia M, Alonso B, Alvarez MJ, Barrientos MJ, Ayan C, Martin Sanchez V. Effects of 2 physiotherapy programs on pain perception, muscular flexibility, and illness impact in women with fibromyalgia: a pilot study. J Manipulative Physiol Ther. 2009 Jan;32(1):84-92. doi: 10.1016/j.jmpt.2008.07.003. PMID 19121466
- [Result] Morey M, Bargay J, Galmes A, Besalduch J. [Plasma cell leukemia]. Sangre (Barc). 1989 Jun;34(3):245. No abstract available. Spanish. PMID 2762987